CLINICAL TRIAL: NCT03739164
Title: Complete Robotic Tampa Associating Microwave Liver Ablation With Portal Vein Ligation
Brief Title: Tampa Associating Microwave Liver Ablation With Portal Vein Ligation for Staged Hepatectomy (TAMLAPS)
Acronym: TAMLAPS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Florida Hospital Tampa Bay Division (Other)
Responsible Party: Sponsor
Other Study IDs: TAMLAPS
Record Dates: First submitted 2018-11-09; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Liver Cancer; Liver Tumor; Hepatocellular Carcinoma; Hilar Cholangiocarcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular; Klatskin Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Years
Biospecimen Retention: Samples With DNA — Samples of healthy tissue pre and post operation will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a study following the outcomes and survival of patients undergoing the TAMLAPS hepatectomy at Florida Hospital Tampa by Dr. Iswanto Sucandy

ELIGIBILITY:
Inclusion Criteria

* Patients scheduled to undergo the TAMLAPS procedure by Dr. Iswanto Sucandy.

Exclusion Criteria:

* Subjects with history of noncompliance.
* Subjects with physical health, substance abuse, or mental health problems that will limit the subject's ability to meet study requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between the ages of 18 and 80 with indication for hepatectomy of >70% liver volume
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2018-07-18 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth of the Future Liver remnant | 2 weeks
  1. Liver growth determined by measuring the kinetic growth rate obtained from pre-operative and post-op stage one CT evaluations of the FLR volume

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Hospital Tampa, Tampa, Florida, United States